CLINICAL TRIAL: NCT06050291
Title: A Study to Assess the Effect of Food on the Bioavailability of Obicetrapib and Ezetimibe After Administration of a Fixed-Dose Combination Formulation of Obicetrapib/Ezetimibe, 10 mg/10 mg in Healthy Adult Subjects
Brief Title: Investigating the Effect of Food on the Bioavailability of a Fixed Dose Combination of Obicetrapib and Ezetimibe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OBEZ-103
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Open-Label, Single-Dose, Randomized, Two-Treatment, Two-Period, Two-Sequence, Crossover Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FDC Tablet Fed + Fast (Experimental): Participants will receive a single Obicetrapib/Ezetimibe, 10 mg/10 mg FDC Tablet in a fed condition on Day 1 of treatment followed by a single Obicetrapib/Ezetimibe, 10 mg/10 mg FDC Table in a fasted condition after, at a minimum, a 56 day washout.
  Interventions: Drug: Fixed-Dose Combination (FDC) Tablet
- FDC Tablet Fast + Fed (Experimental): Participants will receive a single Obicetrapib/Ezetimibe, 10 mg/10 mg FDC Tablet in a fasted condition on Day 1 of treatment followed by a single Obicetrapib/Ezetimibe, 10 mg/10 mg FDC Table in a fed condition after, at a minimum, a 56 day washout.
  Interventions: Drug: Fixed-Dose Combination (FDC) Tablet

INTERVENTIONS:
Drug: Fixed-Dose Combination (FDC) Tablet — Obicetrapib/Ezetimibe FDC tablet

SUMMARY:
This study will assess the effect of food on the bioavailability of obicetrapib and ezetimibe after a single-dose administration of a fixed-dose combination formulation of obicetrapib/ezetimibe, 10 mg/10 mg in healthy adult male and female subjects under fasted and fed conditions.

DETAILED DESCRIPTION:
This is an open-label, single-dose, randomized, two-treatment, two-period, two-sequence crossover relative bioavailability study under fasted and fed conditions. It will assess the effect of food on the bioavailability of obicetrapib and ezetimibe after a single-dose administration of a fixed-dose combination formulation of obicetrapib/ezetimibe, 10 mg/10 mg in healthy adult male and female subjects under fasted and fed conditions. The screening period will be up to 28 days. Patients that are eligible will enter the clinical facility at least 10.5 hours prior to dosing. Depending on their randomization patients will be fed or fasted prior to dosing. They will remain confined for at least 24 hours. After leaving confinement, patients will return to the clinic 9 times for blood draws. At least 56 days after the first dosing, patients will return to the clinic and go through the same process. Those previously fed before dosing will be fasted and those previously fasted will be fed. Patients will return 9 times after their second confinement for additional blood draws.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and Females aged 18 to 65.
* Body Mass Index (BMI) of 18.5-29.9 kg/m², inclusive.
* Females of childbearing potential must be willing to use approved method of birth control.
* Blood pressure 90/60 - 140/90 mmHg, inclusive.
* Hemoglobin level above lower limit of normal.
* Good health.

Key Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.
* History of allergy, sensitivity to obicetrapib, ezetimibe or any components of the study products, or history of any drug hypersensitivity or intolerance that may compromise the safety of the subject.
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction especially hypothyroidism, renal or hepatic disorders, cardiovascular disorders, respiratory disorders, diabetes or obesity.
* Clinically significant history or presence of gastrointestinal disease or history of malabsorption within the last year.
* History of psychiatric disorders occurring within the last two years that required the subject to be hospitalized or treated with medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of statins, cyclosporine, fibrates (e.g., fenofibrate), bile acid seuqstrants (e.g., cholestyramine), or coumarin anticoagulants within 30 days before initial dosing.
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes (especially inducers and inhibitors of CYP3A4) within 30 days before initial dosing.
* Use of any drug that can alter the absorption of other drugs by affecting gastrointestinal motility or by changing the gastric pH, in the opinion of the Investigator, within 14 days before initial dosing.
* Use of any drug that can increase or decrease the metabolism and excretion of the study drug, within 14 days before initial dosing.
* Receipt of any drug as part of a research study within 30 days before initial dosing.
* Previous participation in a research study with obicetrapib.
* Drug or alcohol addiction requiring treatment in the 12 months before initial dosing.
* History of excessive alcohol consumption (on average more than 14 units of alcohol/week) during the past 12 months.
* Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before initial dosing.
* Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* If female, has a positive pregnancy test at screening.
* Use of tobacco- or nicotine-containing products within 30 days before initial dosing.
* Difficulty swallowing tablets or capsules whole.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Cmax | 528.00 hours
  Maximum measured plasma concentration following each treatment.
AUC0-t | 528.00 hours
  Area under the plasma concentration versus time curve from time zero to the time of the last measurable plasma concentration, as calculated by linear trapezoidal method.
AUC0-∞ | 528.00 hours
  Area under the plasma concentration versus time curve from time zero to infinity where AUC0-∞ = AUC0-t + Ct/λz. Ct is the last measurable concentration and λz is the terminal rate constant.

SECONDARY OUTCOMES:
Tmax | 528.00 hours
  Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.
Tlag | 528.00 hours
  Time delay in achieving Tmax
λz | 528.00 hours
  First order rate constant associated with the terminal (log-linear) portion of the curve.
t½ | 528.00 hours
  The terminal half-life will be calculated as ln(2)/λz.
CL/F | 528.00 hours
  Apparent oral systemic clearance, calculated as Dose/AUC0-∞
Vd/F | 528.00 hours
  Apparent volume of distribution during terminal phase, calculated as Dose/(AUC0-∞ × λz)
R2 adjusted | 528.00 hours
  Goodness of fit statistic for the terminal phase, adjusted for the number of points used in the estimation of λz.
AUC_%Extrap_obs | 528.00 hours
  The residual area in percentage will be determined by the formula, [(AUC0-∞-AUC0-t)/AUC0-∞] × 100.

CONTACTS AND LOCATIONS:
Locations (1):
- NOVUM, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No